## Research title

Effects of Tactile Massage in Long-Term Care Facilities

## **NCT** number

NCT05052138

## Date

2021/09/10

## **Abstract**

**Background:** The older residents in the long-term care facilities (LTCFs) frequently suffer from loneliness, anxiety, and depressive symptoms which might affect residents' quality of life and even increase their mortality. Improving residents' psychological health problems is one of the important tasks for nursing staff. There is a need to develop an easy, accessible, and cost-effective intervention in improving older residents' negative emotions. Tactile massage (TM) is a soft touch and through skin-to-skin contact, the oxytocin can be induced to make individual feel relaxed, feel pleasure, and reduce anxiety. Individual might experience a sense of security and feel of being cared for via TM.

**Objective:** To evaluate the effects of tactile massage in improving older residents' psychological health in LTCFs.

**Design:** A randomised controlled trial.

Methods: The randomized controlled trial research design and convenience sampling will be employed. LTCFs will be selected and contacted by researchers. The intervention group received TM for both hands twice a week for four weeks, and the comparison group received regular care. Data were collected before and after the intervention using demographic characteristics information, UCLA Loneliness Scale version 3, Geriatric Anxiety Inventory, Geriatric Depression Scale short form, and Chinese Happiness Scale. In addition, comfort level, relaxation level, and vital signs were also measured before and after each intervention.

Generalized Estimation Equations (GEE) was used to evaluate the effectiveness of the intervention.